CLINICAL TRIAL: NCT04303390
Title: 24 Versus 48 Hours of First Generation or Second Generation Cephalosporin as Prophylaxis to Reduce Surgical Site Infection in Adult Cardiac Surgery Patients: a Randomized Controlled Trial
Brief Title: 24 Vs 48 Hours of Cefazolin or Cefuroxime as Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saud Al Babtain Cardiac Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBCC-2017-14
Record Dates: First submitted 2019-11-03; First posted 2020-03-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefuroxime; Cefazolin

STUDY DESIGN:
Intervention Model Description: 50% of study patients will be assigned to first generation cephalosporin while the other 50% will be assigned to the second generation cephalosporin. 50% of the entire study participants will be assigned to 24 hour therapy while the other 50% will be assigned to 48 hours
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 24 hour Cefuroxime arm (Active Comparator): 25% of the entire study participants are assigned to 24 hours and second generation cephalosporin
  Interventions: Drug: Cefuroxime; Other: 24 hours
- 24 hour Cefazolin arm (Active Comparator): 25% of the entire study participants are assigned to 24 hours and first generation cephalosporin
  Interventions: Drug: Cefazolin; Other: 24 hours
- 48 hour Cefuroxime arm (Active Comparator): 25% of the entire study participants are assigned to 48 hours and second generation cephalosporin
  Interventions: Drug: Cefuroxime; Other: 48 hours
- 48 hour Cefazolin arm (Active Comparator): 25% of the entire study participants are assigned to 48 hours and first generation cephalosporin
  Interventions: Drug: Cefazolin; Other: 48 hours

INTERVENTIONS:
Drug: Cefuroxime — second generation cephalosporin
  Arms: 24 hour Cefuroxime arm; 48 hour Cefuroxime arm
Drug: Cefazolin — First generation cephalosporin
  Arms: 24 hour Cefazolin arm; 48 hour Cefazolin arm
Other: 24 hours — Duration of antibiotic therapy
  Arms: 24 hour Cefazolin arm; 24 hour Cefuroxime arm
Other: 48 hours — Duration of antibiotic therapy
  Arms: 48 hour Cefazolin arm; 48 hour Cefuroxime arm

SUMMARY:
A randomized control trial studying the effect of prophylactic antibiotics to reduce surgical site infections following cardiac surgery in adults using 1st generation cephalosporin (Cefazolin) or 2nd generation cephalosporin (Cefuroxime).

DETAILED DESCRIPTION:
A prospective randomized controlled patient blinded study with 2x2 factional design. It aims to study optimal duration of antibiotic to reduce surgical site infections following cardiac surgery in adults 24 or 48 hours using 1st generation cephalosporin (Cefazolin) or 2nd generation cephalosporin (Cefuroxime). Patients shall remain on either medicines for 24 or 48 hours. The primary endpoints of the study are:(1) 48 hours antibiotic prophylaxis is superior to 24 hours in adult cardiac surgery (2) Cefuroxime is superior to Cafazolin as a prophylactic antibiotic in adult cardiac surgery. Secondary endpoints include; organisms causing surgical site infections, length of hospital and ICU stay, and worsening in renal function.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Planned to undergo a cardiac surgical procedure

Exclusion Criteria:

* Patients on antibiotics on the day of surgery or those who received any within 7 days for any reason
* Patients taken to operating room as salvage
* Patients who are allergic to either cefuroxime or cefazolin
* Patients for LVAD or ECMO
* Patients who are known MRSA carriers
* Patients receiving steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
surgical site infection rate is less with Cefuroxime than Cefazolin | within 3 months from date of surgery
  that Second Generation Cefalosporin is superior to first generation
surgical site infection rate is less with 48 hours rather than 24 hours | within 3 months from date of surgery
  That Longer duration of prophylaxis is better than shorter duration

SECONDARY OUTCOMES:
Length of actual Hospital Stay in the group assigned to 48 hours of cefuroxime | within 3 months from date of surgery
  that 48 hours of cefuroxime will reduce hospital stay
Length of ICU Stay will be shorter in the group assigned to 48 hours of cefuroxime | within 3 months from date of surgery
  that 48 hours of cefuroxime will reduce ICU stay
rate of infection with a specific organism following each of the antibiotics used | within 3 months from date of surgery
  type of organism following each type of antibiotic used
change from baseline of serum creatinine for each antibiotic used | within 3 months from date of surgery
  that 48 hours of cefuroxime will not worsen renal function

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Koudieh, MD, Principal Investigator — Saud AlBabtain Cardiac Center; Shukri M AlSaif, MD, Principal Investigator — Saud AlBabtain Cardiac Center
Locations (1):
- Saud AlBabtain Cardiac Center, Dammam, Eastern Province, Saudi Arabia